CLINICAL TRIAL: NCT00121771
Title: A Phase 1 Trial of the Malaria Candidate Vaccines FP9 CS and MVA CS in Adult Gambian Men Aged 18 - 45 Years
Brief Title: Malaria Candidate Vaccines FP9 Circumsporozoite (CS) and MVA CS in Adult Gambian Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council (Other Government); University of Oxford (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ITDCVG28; VAC 026
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: Malaria; Vaccines; Safety; Immunogenicity
MeSH Terms: conditions — Malaria

INTERVENTIONS:
Biological: FP9 CS
Biological: MVA CS

SUMMARY:
Animal and human studies have shown that the prime-boost immunization strategy using malaria antigens expressed in plasmid or viral vectors induces strong cellular immune responses. An immunization regimen with the malaria vaccines DNA ME-TRAP followed by MVA ME-TRAP induced strong T cell responses in adults in the United Kingdom (UK) and in the Gambia but did not provide significant clinical protection against infection. The investigators assessed two new vaccines which utilize a similar immunization strategy but a different malaria antigen, a circumsporozoite (CS) protein. The entire CS protein was expressed either in a modified vaccinia virus Ankara (MVA) CS, or an attenuated fowlpox virus strain (FP9) CS.

DETAILED DESCRIPTION:
Objectives:

The primary aim was the assessment of safety and reactogenicity of these vaccines in Gambian adults. The secondary aim was the assessment of immunogenicity and comparison with UK adults given the same vaccines.

Study Area:

The study was conducted in the town of Farafenni, about 200km east of the capital city, Banjul. In this area, malaria is highly seasonal with an entomological inoculation rate between 10-50 bites per year. This study was carried out from January to June, when the incidence of malaria is low.

Study Population:

The study involved 32 healthy Gambian adults aged 18-45 years. Volunteers were subjected to a thorough physical and medical examination. Exclusion criteria included a low PCV (< 30%); raised plasma creatinine or ALT levels; and HIV positivity, as determined by ELISA assays.

Study Procedure:

After prior consultations with community leaders, public meetings were held to inform the community of the planned study. Volunteers aged 18-45 years were then invited to take part in the study after written informed consent was obtained in the presence of the principal investigator. Prior to the start of the screening exercise, the investigators checked the age and identity of each volunteer and conducted pre-HIV test counselling. Screening involved a thorough physical examination, blood sampling for haematological (full blood count, packed cell volume [PCV]), renal (plasma creatinine) and hepatic (alanine aminotransferase) tests and HIV 1 and 2 testing by ELISA. All eligible volunteers were issued unique study numbers and photo identification cards.

The initial part of the study was designed to determine the dose and safety of the individual vaccines using an open-label dose escalation method. Study volunteers were randomly allocated to two groups of four that received 5 x 10^7 pfu id of either FP9 CS or MVA CS. When a good safety profile was evident one week after this dose, another set of four volunteers per group received a higher dose (1 x 10^8 pfu id) of FP9 CS or MVA CS. After the investigators had achieved a satisfactory safety profile with a higher dose of both vaccines given alone, they proceeded to administer the vaccines in combination using the heterologous prime-boost regime. The vaccines were administered at 4-week intervals. Eight volunteers received FP9 CS at week 0 followed by MVA CS at week 4 (FM group). Another set of 8 volunteers received FP9 CS at weeks 0 and 4, followed by MVA CS at week 8 (FFM). Following vaccination, volunteers were observed for 1 hour and given a course of antipyretic (paracetamol) to take if required. A physician and a study nurse could be contacted by the volunteers at anytime during the course of the study. In addition, home visits were made by field workers on days 1, 2, 7 and 28, after each vaccination, to record adverse events using a standard questionnaire.

Sample Size:

Sample size was determined by the requirement to make a preliminary evaluation of inter-group and inter-individual variability, to avoid excessive risk and to allow for a realistic workload. Statistical significance may not be reached in this study with low power, but a non-significant finding would provide justification for the need for a study with greater power.

Data Safety Monitoring Board (DSMB):

An international DSMB was established to monitor the conduct of the trial and to approve the analytical plan. The trial was conducted in line with the ICH Good Clinical Practices guidelines and with the Medical Research Council (MRC) rules and regulations for the conduct of clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male aged 18-45 years

Exclusion Criteria:

* Clinically significant history of skin disorder (eczema, psoriasis, etc.), allergy, immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease or neurological illness
* Any clinical evidence of immunosuppression such as oral candida, stomatitis, aphthous or septic ulceration, septic skin lesions or any clinical or laboratory evidence of infection or immunocompromise
* History of splenectomy
* Haematocrit of less than 30%
* Serum creatinine concentration >130mmol/L
* Serum ALT concentration >42IU/L
* Blood transfusion within one month of the beginning of the study
* Administration of any other vaccine or immunoglobulin within two weeks before scheduled MVA vaccination
* Positive HIV antibody test
* Current participation in another clinical trial, or within 12 weeks of this study
* Any other finding which, in the opinion of the investigators, would increase the risk of an adverse outcome from participation in the trial
* Likelihood of travel away from the study area for the duration of the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32
Dates: Start 2004-01; Study Completion 2004-07

PRIMARY OUTCOMES:
Safety and immunogenicity

SECONDARY OUTCOMES:
Comparison of immunogenicity with non-immune UK adults

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, MD, Phd, Study Chair — Centre for Human Genetics, University of Oxford
Locations (1):
- Medical Research Council Laboratories, Banjul, The Gambia